CLINICAL TRIAL: NCT03929367
Title: Pharmacokinetics of Intravenous Oxytocin and Effects on Sensory Function in Healthy Volunteers
Brief Title: PK Sampling After IV Oxytocin and Effects on Sensory Function in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00056413
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Results first posted 2021-04-19 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Single intravenous administration of oxytocin (Pitocin®), 10 IU
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Oxytocin (Pitocin®), 10 IU (Other): Oxytocin 10 IU administered once per intravenous injection
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Single IV administration of oxytocin
  Other Names: Pitocin

SUMMARY:
The primary goal of this protocol is to model change in oxytocin concentrations in plasma after intravenous (IV) administration. Additional measurements will be performed on sensory function that could be influenced by oxytocin during later time periods when blood samples are widely separated by time. This protocol will describe the pharmacokinetics (PK) of intravenous oxytocin in healthy adult men and adult,non-pregnant women. PK samples will be obtained after an injection of intravenous oxytocin 10 IU over 60 seconds.

Blood will be drawn for the PK samples prior to the oxytocin administration and then 11 times after administration.

There are two additional measures which will assess two different aspects of sensory function.

MEASURE 1: Light Touch Frequency Threshold In order to determine the highest frequency that specific nerve fibers can respond to, a simple device that produces an oscillatory / vibratory stimulus will be used on the hand. The subject places fingertips, palm, and palm side of the wrist sequentially and the device is set to slowly decrease the frequency of vibration from 1 kHz until the subject first perceives this. This is repeated three times at each site and takes less than 5 minutes in total. This will be performed before the oxytocin administration and 6 times after the administration of IV Oxytocin.

MEASURE 2: Sustained Heat The surface of the skin of the forearm or leg is heated to 113°F using a computer controlled thermode for a period of 5 minutes. This will be done before the IV Oxytocin and 4 times after the administration. A set of random thermal temperatures (98°F-122°F) will also be applied to the skin of the leg or forearm before the IV Oxytocin administration and 4 times after administration of IV Oxytocin.

DETAILED DESCRIPTION:
The primary goal of this protocol is to model change in oxytocin concentrations in plasma after intravenous administration, (oxytocin (Pitocin®), 10 IU) the investigators will also acquire tests of sensory function that could be modulated by oxytocin during later time periods when blood samples are widely separated by time. There are two measures which will assess two different aspects of sensory function.

MEASURE 1: Light Touch Frequency Threshold Light touch is subserved by a group of myelinated peripheral nerves with fast conduction in the Aβ range and which are capable of following high frequencies, being responsible for the sensation of vibration. This capability of individual nerve fibers to respond with high frequency also underlies our ability to sense a light touch moving across the body surface as in brushing.

In preclinical studies investigators have shown that, following injury, these light touch fibers lose their ability to follow high frequencies and, in some cases, no longer respond to mechanical stimulation at all. Oxytocin, when perfused around the neuronal cell bodies of these Aβ nerve fibers, partially restores their function, including their response to high frequency stimulation.

In order to determine the highest frequency that Aβ nerve fibers can respond to, the investigators have created a simple device that produces an oscillatory / vibratory stimulus which can be used on the hand. The subject places fingertips, palm, and volar aspect of the wrist sequentially and the device is set to slowly decrease the frequency of vibration from 1 kilohertz (kHz) until the participant first perceives this. This is repeated three times at each site and takes under 5 minutes in total.

The investigators anticipate that oxytocin will have no effect on normal Aβ fibers and that this measure will not change after oxytocin administration. This will provide important data to contrast with the expected efficacy of oxytocin in the setting of injury, to be studied in subsequent protocols.

MEASURE 2: Sustained Heat As part of a protocol used by the investigators in several studies, the surface of the skin of the forearm or leg is heated to 45°C using a computer-controlled thermode for a period of 5 minutes. This typically results in a slowly increasing pain experience, peaking at 5 minutes in the mild to low moderate range and has been tolerated by more than 150 subjects in studies over the past 14 years.

In an interim analysis of an ongoing clinical study in volunteers, the investigators noted that spinal injection of oxytocin, 15 μg (equivalent to 9 IU), that pain from this sustained heat was dramatically reduced over the 5 minutes of stimulus presentation. In contrast, spinal oxytocin had no effect on the stimulus-response relationship of pain to noxious heat over a 42-50°C range when the stimuli were presented for only 5 seconds. These data suggest that oxytocin reduces C-fiber mediated signaling of sustained heat pain, likely through a spinal site of action.

Drugs administered spinally have a much higher concentration in cerebrospinal fluid than plasma. Nonetheless, spinally administered drugs are typically absorbed to an extent and with a time course similar to that after intramuscular injection, and it is conceivable that the effect on sustained heat pain investigators are seeing in the spinal study reflect peripheral effects via systemic absorption. Thus, if the investigators see a similar reduction in response to sustained heat in this protocol of intravenous administration, the investigators will conclude that oxytocin is more likely activating peripherally than spinally.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 and < 60 years of age, Body Mass Index (BMI) <40.
* Generally in good health as determined by the Principal Investigator based on prior medical history, American Society of Anesthesiologists physical status I or II
* Normal blood pressure (systolic 90-140 mmHg; diastolic 50-90 mmHg) resting heart rate 45-100 beats per minute) without medication
* Female subjects of child-bearing potential and those < 1 year post-menopausal, must be practicing highly effective methods of birth control such as hormonal methods

Exclusion Criteria:

* Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
* Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
* Women who are pregnant (positive result for serum pregnancy test at screening visit), women who are currently nursing or lactating, women that have been pregnant within 2 years
* Subjects with neuropathy, chronic pain, diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shafer SL, Ririe DG, Miller S, Curry RS, Hsu DT, Sullivan GM, Eisenach JC. Plasma pharmacokinetics of intravenous and intranasal oxytocin in nonpregnant adults. Br J Anaesth. 2025 May;134(5):1513-1522. doi: 10.1016/j.bja.2024.12.046. Epub 2025 Mar 21. PMID 40121179

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: None. All enrolled subjects completed the study.
Period: Overall Study
Arm/Group | Oxytocin (Pitocin®), 10 IU
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 29 (3.4)
Height [Mean (Standard Deviation); unit: cm] | 173 (6.5)
Weight [Mean (Standard Deviation); unit: kg] | 86 (11)
Light Touch Frequency Threshold [Mean (Standard Deviation); unit: Hz] — The frequency at which the vibration is perceived before intravenous oxytocin administration
  Hz | 731 (155)
Sustained heat [Mean (Standard Deviation); unit: units on a scale] — 0-10 verbal pain score to a 45 degree Celsius stimulus before intravenous oxytocin administration; higher score denotes worse outcome. Population: Technical failure in one subject, leaving only 10 evaluable
  units on a scale
    One minute: number analyzed (Participants) | 10
    One minute | .36 (.21)
    Two minutes: number analyzed (Participants) | 10
    Two minutes | .68 (.32)
    Three minutes: number analyzed (Participants) | 10
    Three minutes | .64 (.29)
    Four minutes | .82 (.25)
    Five minutes: number analyzed (Participants) | 10
    Five minutes | 1.32 (.3)

OUTCOME MEASURES:

1. Primary Outcome: Oxytocin Concentration
Description: Plasma concentrations of oxytocin at defined times after intravenous infusion
Time Frame: 2 minutes
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
pg/ml | 1047 (556)
Statistical Analysis 1: Comparison: Oxytocin (Pitocin®), 10 IU; Test type: Other — Modeling of change of plasma oxytocin concentration over time using nonlinear canonical compartment model; Bayesian information criterion = 2

2. Primary Outcome: Oxytocin Concentration
Description: Plasma concentrations of oxytocin at defined times after intravenous infusion
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
pg/ml | 587 (257)

3. Primary Outcome: Oxytocin Concentration
Description: Plasma concentrations of oxytocin at defined times after intravenous infusion
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
pg/ml | 322 (136)

4. Primary Outcome: Oxytocin Concentration
Description: Plasma concentrations of oxytocin at defined times after intravenous infusion
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
pg/ml | 202 (91)

5. Primary Outcome: Oxytocin Concentration
Description: Plasma concentrations of oxytocin at defined times after intravenous infusion
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
pg/ml | 82 (40)

6. Primary Outcome: Oxytocin Concentration
Description: Plasma concentrations of oxytocin at defined times after intravenous infusion
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
pg/ml | 41 (20)

7. Primary Outcome: Oxytocin Concentration
Description: Plasma concentrations of oxytocin at defined times after intravenous infusion
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
pg/ml | 25 (13)

8. Primary Outcome: Oxytocin Concentration
Description: Plasma concentrations of oxytocin at defined times after intravenous infusion
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
pg/ml | 10 (5.6)

9. Primary Outcome: Oxytocin Concentration
Description: Plasma concentrations of oxytocin at defined times after intravenous infusion
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
pg/ml | 6.2 (3.6)

10. Primary Outcome: Oxytocin Concentration
Description: Plasma concentrations of oxytocin at defined times after intravenous infusion
Time Frame: 180 minutes
Population: In 7 subjects oxytocin concentration was below the limit of detection (1 pg/ml)
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 4
pg/ml | 2.5 (1.6)

11. Primary Outcome: Oxytocin Concentration
Description: Plasma concentrations of oxytocin at defined times after intravenous infusion
Time Frame: 240 minutes
Population: In 9 subjects oxytocin concentration was below the limit of detection (1 pg/ml)
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 2
pg/ml | 1.0 (1.5)

12. Secondary Outcome: Light Touch Frequency Threshold
Description: The frequency at which the vibration is perceived after intravenous oxytocin administration
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
Hz | 722 (141)
Statistical Analysis 1: Comparison: Oxytocin (Pitocin®), 10 IU; Test type: Superiority — Light touch detection frequency was compared over time in comparison to baseline using a one way analysis of variance for repeated measures. A power analysis was not performed for this secondary outcome measure; p = .89, ANOVA — No effect

13. Secondary Outcome: Light Touch Frequency Threshold
Description: The frequency at which the vibration is perceived after intravenous oxytocin administration
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
Hz | 710 (130)

14. Secondary Outcome: Light Touch Frequency Threshold
Description: The frequency at which the vibration is perceived after intravenous oxytocin administration
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
Hz | 732 (128)

15. Secondary Outcome: Light Touch Frequency Threshold
Description: The frequency at which the vibration is perceived after intravenous oxytocin administration
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
Hz | 727 (127)

16. Secondary Outcome: Light Touch Frequency Threshold
Description: The frequency at which the vibration is perceived after intravenous oxytocin administration
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
Hz | 693 (154)

17. Secondary Outcome: Light Touch Frequency Threshold
Description: The frequency at which the vibration is perceived after intravenous oxytocin administration
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 11
Hz | 771 (99)

18. Secondary Outcome: Sustained Heat
Description: 0-10 verbal pain score to a 45 degree Celsius stimulus after intravenous oxytocin administration; higher score denotes worse outcome.
Time Frame: 31 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | 0.36 (.21)

19. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 32 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .14 (.14)
Statistical Analysis 1: Comparison: Oxytocin (Pitocin®), 10 IU; Test type: Superiority — Sustained heat score at the end of each 5 minute session was compared to baseline across time using a one-way analysis of variance for repeated measures. Power analysis was not performed for this secondary outcome measure; p = 0.014, ANOVA

20. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 33 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .32 (.2)

21. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 34 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .32 (.2)

22. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 35 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .64 (.29)

23. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 61 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .45 (.33)

24. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 62 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .23 (.13)

25. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 63 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .27 (.15)

26. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 64 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .36 (.16)

27. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 65 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .73 (.25)

28. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 121 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .36 (.21)

29. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 122 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .23 (.13)

30. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 123 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .18 (.19)

31. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 124 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .27 (.2)

32. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 125 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .77 (.37)

33. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 181 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .27 (.2)

34. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 182 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .18 (.13)

35. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 183 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .32 (.15)

36. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 184 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .59 (.21)

37. Secondary Outcome: Sustained Heat
Description: as for outcome 18
Time Frame: 185 minutes
Population: Technical failure in one subject, leaving 10 evaluable
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin (Pitocin®), 10 IU
Number analyzed (Participants) | 10
score on a scale | .86 (.22)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Oxytocin (Pitocin®), 10 IU: This was a one day, open-label, single-dose study of intravenous oxytocin for the purpose of estimating plasma pharmacokinetic model parameters in adult men and women. Blood pressure, heart and respiratory rate, and oxyhemoglobin saturation were recorded prior to and at intervals following administration of oxytocin. In addition, subjects were informed to indicate if they had any subjective symptoms.
Arm/Group | Oxytocin (Pitocin®), 10 IU
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (Pitocin®), 10 IU (N=11)
Facial flushing (Cardiac disorders) | 7 (7) — Sensation of facial flushing lasting 2-12 minutes without visual appearance of flushing
Headache (Nervous system disorders) | 3 (3) — Mild headache lasting 2-12 min after oxytocin administration
Increased heart rate (Cardiac disorders) | 3 (3) — Sensation of increased heart rate or heart pounding, but not accompanied by tachycardia or hypertension by direct measurement

LIMITATIONS AND CAVEATS:
Technical failure in one individual resulting in uninterpretable pain scores to sustained heat as a secondary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT03929367/Prot_SAP_001.pdf
  • Informed Consent Form (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT03929367/ICF_000.pdf